CLINICAL TRIAL: NCT07057739
Title: Fentanyl and Dexmedetomidine as Adjuvants to Bupivacaine in Ultrasound-guided Superficial Cervical Plexus Block in Thyroid Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Adel Abd Elmoaty Basyouni Elabd, Resident at Anaesthesia, Surgical Intensive Care and Pain Management , Faculty of Medicine, Kafr Elsheikh University Kafr Elsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-186
Record Dates: First submitted 2025-06-17; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Fentanyl; Dexmedetomidine; Adjuvants; Bupivacaine; Ultrasound; Superficial Cervical Plexus Block; Thyroid Surgeries
MeSH Terms: interventions — Bupivacaine; Sodium Chloride; Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Control) (Experimental): Patients received superficial cervical plexus block with 1 ml of normal saline with 7ml bupivacaine 0.25% per side without adjuvants.
  Interventions: Drug: Superficial cervical plexus block
- Group F (Fentanyl) (Experimental): Patients received superficial cervical plexus block with fentanyl 1 ml (50 microgram) as an adjuvant to 7ml bupivacaine 0.25% per side.
  Interventions: Drug: Superficial cervical plexus block + Fentanyl
- Group D (Dexmedetomidine) (Experimental): Patients received superficial cervical plexus block with dexmedetomidine 0.5mcg/kg in 1 ml of normal saline as an adjuvant to 7ml bupivacaine 0.25% per side.
  Interventions: Drug: Superficial cervical plexus block + Dexmedetomidine

INTERVENTIONS:
Drug: Superficial cervical plexus block — Patients received superficial cervical plexus block with 1 ml of normal saline with 7ml bupivacaine 0.25% per side without adjuvants.
  Other Names: Bupivacaine 0.25% + Saline
  Arms: Group C (Control)
Drug: Superficial cervical plexus block + Fentanyl — Patients received superficial cervical plexus block with fentanyl 1 ml (50 microgram) as an adjuvant to 7ml bupivacaine 0.25% per side.
  Other Names: Bupivacaine 0.25% + Fentanyl
  Arms: Group F (Fentanyl)
Drug: Superficial cervical plexus block + Dexmedetomidine — Patients received superficial cervical plexus block with dexmedetomidine 0.5mcg/kg in 1 ml of normal saline as an adjuvant to 7ml bupivacaine 0.25% per side.
  Other Names: Bupivacaine 0.25% + Dexmedetomidine
  Arms: Group D (Dexmedetomidine)

SUMMARY:
This study aimed to compare the analgesic efficacy between fentanyl and dexmedetomidine as adjuvants to bupivacaine in ultrasound-guided superficial cervical plexus block for thyroid surgeries.

DETAILED DESCRIPTION:
Cervical plexus blocks are easy to perform and provide anesthesia for the surgical procedure in the distribution of C2 to C4, including carotid endarterectomies, lymph node dissection, and thyroid surgeries.

Dexmedetomidine (α2 adrenoceptor agonist) is being used for intravenous (IV) sedation and analgesia for intubated and mechanically ventilated patients in Intensive Care Units. Its use in peripheral nerve blocks has recently been described. It has been reported to have a rapid onset time,prolong the duration of local anesthetics, and it is approximately 8 times more potent than clonidine and is also reportedly safe and effective in peripheral nerve blocks.

Opiates are widely known to have an analgesic effect at the central and spinal cord level. However, opioid analgesia can be initiated by activation of peripheral opioid receptors. Opioids such as fentanyl have been used for regional nerve plexus blocks to improve the block duration and quality.

ELIGIBILITY:
Inclusion Criteria:

* Patient's approval.
* Aged 20-65 years
* American Society of Anesthesiologists (ASA) physical status I or II
* Undergoing thyroid surgery
* Euthyroid patients

Exclusion Criteria:

* Patient refusal.
* Age: >65 and <20 years.
* Allergy to Dexmedetomidine, local anesthetics, systemic opioids and any of the drugs included in the multimodal perioperative pain protocol.
* Patient with coagulation disorders.
* Chronic pain syndromes and patients with chronic opioid use are defined as use of regular daily doses of systemic narcotics for the past 6 months prior to the surgery.
* BMI of 35 kg/m2 or more.
* Physical Status: American Society of Anesthesiologists (ASA) III & IV.
* Local infection or sepsis at the site of injection.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Pain degree | 24 hours postoperatively
  Postoperative pain was assessed using a 10-point Visual Analog Scale (VAS), where 0 represents no pain and 10 indicates the worst imaginable pain. It was assessed at 0, 2, 4, 6, 8, 12, 18, and 24 hours post-surgery.

SECONDARY OUTCOMES:
Duration of Sensory Block | 24 hours postoperatively
  Time from performance of the superficial cervical plexus block to the complete resolution of sensory blockade was assessed.
Time to First Rescue Analgesia | 48 hours postoperatively
  Time from end of surgery to the administration of the first dose of rescue analgesia, triggered by VAS score ≥3.
Total Opioid Consumption | 48 hours postoperatively
  Cumulative dose of opioid analgesics (pethidine in mg) administered during the first 48 hours postoperatively.
Mean arterial pressure (MAP) | 24 hours postoperatively
  Serial measurement of mean arterial pressure (MAP, mmHg) at baseline, intraoperatively every 30 minutes, and postoperatively at 0, 2, 4, 6, 8, 12, and 24 hours.
Heart rate | 24 hours postoperatively
  Serial measurement of heart rate (beats per minute) at baseline, intraoperatively every 30 minutes, and postoperatively at 0, 2, 4, 6, 8, 12, and 24 hours.
Incidence of Adverse Events | 48 hours postoperatively
  Incidence of adverse events including but not limited to Horner's syndrome, local anesthetic systemic toxicity (LAST), phrenic nerve block, bradycardia, hypotension, hematoma, nausea, vomiting, respiratory discomfort, and failed block was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr Elsheikh University, Kafr ash Shaykh, Kafr Elsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.